CLINICAL TRIAL: NCT04332926
Title: Effects of E-Cigarette Nicotine Content in Smokers (Nicotine Flux Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HM20018290; 2U54DA036105 (NIH)
Record Dates: First submitted 2020-03-25; First posted 2020-04-03 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Electronic Cigarette Use
Keywords: Electronic Cigarette; Nicotine Flux
MeSH Terms: conditions — Vaping | interventions — Restraint, Physical; Nicotine

STUDY DESIGN:
Masking Description: Participants will be blinded to their condition (nicotine level) used in each session, except during their 'own brand' session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Tobacco product administration and assessment, own brand cigarettes; Other: Tobacco product administration and assessment, ECIG 30 Watts, 0 mg/ml nicotine; Other: Tobacco product administration and assessment, ECIG 30 Watts, 8 mg/ml nicotine; Other: Tobacco product administration and assessment, ECIG 30 Watts, 15 mg/ml nicotine; Other: Tobacco product administration and assessment, ECIG 30 Watts, 30 mg/ml nicotine

INTERVENTIONS:
Other: Tobacco product administration and assessment, own brand cigarettes — 4 sample puffs, followed by a 60 minute rest period, hypothetical drug purchase tasks, followed by progressive ratio tasks (single product and two products, with 60 minute rest in between) where participants work to earn puffs of tobacco products; preceded and followed by physiological and subjective assessment
Other: Tobacco product administration and assessment, ECIG 30 Watts, 0 mg/ml nicotine — 4 sample puffs, followed by a 60 minute rest period, hypothetical drug purchase tasks, followed by progressive ratio tasks (single product and two products, with 60 minute rest in between) where participants work to earn puffs of tobacco products; preceded and followed by physiological and subjective assessment
Other: Tobacco product administration and assessment, ECIG 30 Watts, 8 mg/ml nicotine — 4 sample puffs, followed by a 60 minute rest period, hypothetical drug purchase tasks, followed by progressive ratio tasks (single product and two products, with 60 minute rest in between) where participants work to earn puffs of tobacco products; preceded and followed by physiological and subjective assessment
Other: Tobacco product administration and assessment, ECIG 30 Watts, 15 mg/ml nicotine — 4 sample puffs, followed by a 60 minute rest period, hypothetical drug purchase tasks, followed by progressive ratio tasks (single product and two products, with 60 minute rest in between) where participants work to earn puffs of tobacco products; preceded and followed by physiological and subjective assessment
Other: Tobacco product administration and assessment, ECIG 30 Watts, 30 mg/ml nicotine — 4 sample puffs, followed by a 60 minute rest period, hypothetical drug purchase tasks, followed by progressive ratio tasks (single product and two products, with 60 minute rest in between) where participants work to earn puffs of tobacco products; preceded and followed by physiological and subjective assessment

SUMMARY:
This study aims to better understand how e-cigarettes (ECIG) nicotine flux impacts several behavioral economic measures of abuse liability.

ELIGIBILITY:
Inclusion Criteria:

* healthy (determined by self-report)
* between the ages of 18-55
* willing to provide informed consent
* able to attend the lab and abstain from tobacco/nicotine as required and must agree to use designated products according to study protocol

Exclusion Criteria:

* Women if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening.
* Some study details about the eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline O Cobb, PhD, Principal Investigator — Virginia Commonwealth University; Andrew Barnes, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Center for the Study of Tobacco Products, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Enrollment: When I try to add the individual numbers for the different procedures, it confuses the system since it looks like each procedure is a seperate arm. For feasibility issues the study design was altered from a crossover study to a single-arm parallel one. So for this arm, Tobacco product administration and assessment: 4 sample puffs, followed by a 60 minute rest period, hypothetical drug purchase tasks, followed by progressive ratio tasks (single product and two products, with 60 minute rest in between) where participants work to earn puffs of tobacco products; preceded and followed by physiological and subjective assessment
Period: Overall Study
Arm/Group | Overall Enrollment
Started | 44
Active Comparator: Own Brand Cig | 32 (32 subjects participated in this arm, and 32 completed the arm)
Experimental: ECIG 30 W, 0 mg/ml Nic | 35 (37 subjects participated in this arm, and 35 completed the arm)
Experimental: ECIG 30 W, 8 mg/ml Nic | 34 (35 subjects participated in this arm, and 34 completed the arm)
Experimental: ECIG 30 W, 15 mg/ml Nic | 34 (36 subjects participated in this arm, and 34 completed the arm)
Experimental: ECIG 30 W, 30 mg/ml Nic | 36 (36 subjects participated in this arm, and 36 completed the arm)
Completed | 32
Not Completed | 12
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Tobacco product administration and assessment: 4 sample puffs, followed by a 60 minute rest period, hypothetical drug purchase tasks, followed by progressive ratio tasks (single product and two products, with 60 minute rest in between) where participants work to earn puffs of tobacco products; preceded and followed by physiological and subjective assessment
Arm/Group | Experimental
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.61 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 14
  More than one race | 3
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Effort for Product Puffs With Cross Product Progressive Ratio Task (CP-PRT)
Description: This is now a single-arm parallel study design. The main outcome of interest in the CP-PRT is the relative reinforcing value - defined as how hard a participant is willing to work for the session product compared to their own brand cigarette. The breakpoint, or highest trial number that a participant completed for a puff of the session-specific product will be used as the measure of relative reinforcing value.
Time Frame: The CP-PRT is completed once per study session (except it is not completed in the 5th, own brand session), at 185 minutes into the session.
Population: The study morphed from a cross-over study into a single-arm study due to feasibility issues. Instead of different arms completing the interventions in a different order, all of the subjects were moved into one arm and completed the interventions in the same order.
Measure: Mean (Standard Deviation); unit: Breakpoint (highest trial completed)
Arm/Group | Experimental
Number analyzed (Participants) | 32
Breakpoint (highest trial completed)
  ECIG 30 Watts, 0 mg/ml nicotine | 6.30 (2.83)
  ECIG 30 Watts, 8 mg/ml nicotine | 6.38 (2.94)
  ECIG 30 Watts, 15 mg/ml nicotine | 6.34 (2.70)
  ECIG 30 Watts, 30 mg/ml nicotine | 5.94 (2.93)

2. Primary Outcome: Breakpoint of Drug Purchase Task (DPT)
Description: The DPTs will yield measures of willingness to pay (demand) for session-specific tobacco products. Choices made during this task are not reinforced during the session. Using the DPT, participants estimate the number of session-specific product puffs they would take across increasing prices per puff. DPT demand will be characterized by the Breakpoint (BP); i.e., the highest price per puff at which participants indicate they would stop using the session-specific product rather than incur the cost.
Time Frame: Each DPT will be completed once per study session, about 75 minutes into the session. The results will reported in US dollars ($).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: US dollars ($)
Groups:
- Experimental: For feasibility issues the study design was altered from a crossover study to a single-arm parallel one. So for this arm, Tobacco product administration and assessment: 4 sample puffs, followed by a 60 minute rest period, hypothetical drug purchase tasks, followed by progressive ratio tasks (single product and two products, with 60 minute rest in between) where participants work to earn puffs of tobacco products; preceded and followed by physiological and subjective assessment
Arm/Group | Experimental
Number analyzed (Participants) | 32
US dollars ($)
  Own Brand Cigarette: number analyzed (Participants) | 30
  Own Brand Cigarette | 1.23 (2.10)
  ECIG 30 Watts, 0 mg/ml nicotine | 0.54 (0.90)
  ECIG 30 Watts, 8 mg/ml nicotine | 0.96 (1.78)
  ECIG 30 Watts, 15 mg/ml nicotine: number analyzed (Participants) | 31
  ECIG 30 Watts, 15 mg/ml nicotine | 0.43 (0.77)
  ECIG 30 Watts, 30 mg/ml nicotine | 0.49 (1.01)

3. Primary Outcome: Effort for Product Puffs With Progressive Ratio Task (PRT)
Description: The PRT will yield a measure of willingness to work for session-specific tobacco products (via number of times a space bar is pressed to earn puffs) through the outcome measure: mean number of puffs self-administrated. The outcome measure of interest is the total number of puffs self-administered.
Time Frame: The PRT is completed once per study session, at 85 minutes into the session.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of puffs
Arm/Group | Experimental
Number analyzed (Participants) | 32
Number of puffs
  Own Brand Cigarette | 9.06 (2.73)
  ECIG 30 Watts, 0 mg/ml nicotine | 7.69 (3.51)
  ECIG 30 Watts, 8 mg/ml nicotine | 7.88 (3.42)
  ECIG 30 Watts, 15 mg/ml nicotine | 7.31 (3.89)
  ECIG 30 Watts, 30 mg/ml nicotine | 6.34 (4.37)

ADVERSE EVENTS:
Time Frame: Data were collected during laboratory visits, approximately over 3 weeks; no follow up adverse event data collection occurred.
Description: Non-systematic. Questionnaire assessed at the beginning of each laboratory session, participant self-report. For adverse events that happened outside of the laboratory, no experimental condition is applicable. For adverse events that happened within the laboratory (e.g., during an experimental session), events are reported separately for each relevant experimental condition.
Groups:
- Experimental: The study was originally organized as a cross-over study but due to feasibility circumstances, the study team determined that it was more important to preserve the subject enrollment numbers and complete the study in the most efficient manner for the enrolled subjects. So this became a single-arm parallel study. The study involved Tobacco product administration and assessment: 1) Effort for Product Puffs With Cross Product Progressive Ratio Task (CP-PRT), 2) Breakpoint of Drug Purchase Task (DPT), and 3) Effort for Product Puffs With Progressive Ratio Task (PRT)
  The individual interventions are listed in the milestones section.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 1/44
Other Adverse Events (participants affected / at risk) | 3/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=44)
Surgical and medical procedures: unrelated hysterectomy (Surgical and medical procedures) | 1 (1) — Surgical and medical procedures: unrelated hysterectomy. (Note: adverse event occurred outside of the laboratory; therefore, reporting by experimental condition is not applicable.)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=44)
Elevated Blood Pressure, ECIG 30 W, 30 mg/ml nicotine condition (Blood and lymphatic system disorders) | 3 (3) — Blood pressure was elevated in the ECIG 30 W, 30 mg/ml nicotine condition

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT04332926/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT04332926/ICF_002.pdf